CLINICAL TRIAL: NCT04239911
Title: Leveraging Home Health Aides to Improve Outcomes in Heart Failure: A Pilot Randomized Controlled Trial
Brief Title: Leveraging Home Health Aides to Improve Outcomes in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 19-08020553; K23HL150160-01 (NIH)
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure; Congestive Heart Failure
Keywords: home health aides; home health care; home care agency
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: 104 home health aides will be recruited from VNS Health and randomized to either enhanced usual care arm (heart failure training course; n = 52) or the intervention (heart failure training course plus mHealth app; n =52). Four nurses will also be recruited to the study. The total duration of each home health aides' involvement will be 90 days.
Who Masked: Outcomes Assessor
Masking Description: Data analyst will be blinded to study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced usual care (Active Comparator): Home health aides in the enhanced usual care arm will receive a virtual heart failure training course.
  Interventions: Behavioral: Virtual training course
- Intervention arm (Experimental): Home health aides in the intervention arm will receive a virtual heart failure training course and a communication-based messaging app.
  Interventions: Behavioral: mHealth app; Behavioral: Virtual training course

INTERVENTIONS:
Behavioral: mHealth app — The mHealth app will provide heart failure-specific education to home health aides and allow them to report clinical observations and ask nurses questions in real-time.
  Arms: Intervention arm
Behavioral: Virtual training course — Virtual training course on heart failure for home health aides.

SUMMARY:
The purpose of the study is to determine the effectiveness of an intervention among home health aides caring for adults admitted to home care with a primary diagnosis of heart failure at VNS Health Partners in Care (home care agency). The study will examine the interventions' effect on home health aides' heart failure knowledge and confidence caring for adults with heart failure, as well as on the client's overall health (visits to the emergency department and hospital readmissions).

DETAILED DESCRIPTION:
The investigator's central hypothesis is that an intervention that can optimize and improve the experience of home health aides caring for the heart failure patients has the potential to improve home health aides' own self-efficacy, heart failure knowledge, and also patient outcomes. The intervention for home health aides is comprised of a) remote classroom education on heart failure and b) an mHealth app containing HF educational content and a messaging application that connects HHAs and their nurse supervisors. This intervention requires feasibility and acceptability testing, as well as preliminary testing of its effectiveness among home health aides caring for community-dwelling adults with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Home health aide employed at VNS Health Partners in Care home care agency.
* 1 or more years of experience as a home health aide.
* Speak English or Spanish.
* Assigned to care for an adult admitted to home care with a primary diagnosis of heart failure.

Exclusion Criteria:

* Doesn't meet inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2024-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madeline R Sterling, MD, MPH, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- VNS Health Partners in Care, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sterling MR, Espinosa CG, Vergez S, McDonald MV, Ringel J, Tobin JN, Banerjee S, Dell N, Kern LM, Safford MM. Home Health Aides Caring for Adults With Heart Failure: A Pilot Randomized Clinical Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2548121. doi: 10.1001/jamanetworkopen.2025.48121. PMID 41213039
- [Derived] Espinosa CG, Vergez S, McDonald MV, Safford MM, Cho J, Tobin JN, Mourad O, Marcus R, Joanna Bryan Ringel J, Banerjee S, Dell N, Feldman P, Sterling MR. Leveraging home health aides to improve outcomes in heart failure: A pilot study protocol. Contemp Clin Trials. 2024 Aug;143:107570. doi: 10.1016/j.cct.2024.107570. Epub 2024 May 11. PMID 38740297

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enhanced Usual Care | Intervention Arm
Started | 52 | 53
Completed | 50 | 52
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: Of the 105 participants that consented to be in the study, 3 participants were lost to follow-up between consents and taking the baseline survey.
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care | Intervention Arm | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (10.9) | 54.8 (10.2) | 54.0 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 50 | 98
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 30 | 32 | 62
  American Indian/Alaskan Native | 1 | 0 | 1
  Asian | 3 | 4 | 7
  White | 6 | 3 | 9
  Other | 9 | 12 | 21
  Missing Information on Race | 1 | 1 | 2
Education [Count of Participants; unit: Participants]
  No Degree or Some High School | 9 | 12 | 21
  Completed High School or GED | 18 | 18 | 36
  Some College | 12 | 8 | 20
  College Degree | 8 | 9 | 17
  Graduate Degree | 2 | 5 | 7
  Missing Information on Education | 1 | 0 | 1
Foreign-Born [Count of Participants; unit: Participants]
  Foreign-Born | 45 | 43 | 88
  US-Born | 5 | 9 | 14
Primary Language [Count of Participants; unit: Participants]
  English | 33 | 32 | 65
  Spanish | 11 | 9 | 20
  Other | 6 | 11 | 17
Years as Home Health Aide [Count of Participants; unit: Participants]
  0-5 years | 13 | 15 | 28
  6-10 years | 14 | 17 | 31
  11-15 years | 9 | 7 | 16
  >15 years | 14 | 13 | 27
Number of Home Care Agencies worked for in the past [Count of Participants; unit: Participants]
  0-1 agency | 26 | 27 | 53
  2 agencies | 17 | 16 | 33
  greater than or equal to 3 agencies | 7 | 9 | 16
Years worked at their current agency [Count of Participants; unit: Participants]
  0-5 years | 16 | 19 | 35
  6-10 years | 16 | 18 | 34
  11-15 years | 10 | 8 | 18
  greater than 15 years | 8 | 6 | 14
  Missing Information | 0 | 1 | 1
Number of Heart Failure Patients Cared for [Count of Participants; unit: Participants]
  less than or equal to 5 Heart Failure Patients | 38 | 27 | 65
  greater than 5 Heart Failure Patients | 6 | 12 | 18
  not sure | 6 | 13 | 19
Hours per week spent with Heart Failure client [Count of Participants; unit: Participants]
  1-5 hours per week | 9 | 6 | 15
  6-10 hours per week | 14 | 20 | 34
  11-20 hours per week | 6 | 6 | 12
  Greater than 20 hours per week | 16 | 9 | 25
  Not Sure | 4 | 10 | 14
  Missing Information | 1 | 1 | 2
Heart Failure Training [Count of Participants; unit: Participants]
  None | 24 | 22 | 46
  A little | 13 | 18 | 31
  Some | 13 | 10 | 23
  A lot | 0 | 2 | 2
Management (CC SCHFI) [Median (Inter-Quartile Range); unit: units on a scale] — Management is a subscale of the Caregiver Contribution to Self-Care in HF Index (CC SCHFI). The CC-SCHFI is a 22-item scale which measures caregivers' contributions to: HF maintenance, HF management, and HF caregiving self-efficacy (confidence). The management sub-scale ranges from 0-100. Higher scores indicate higher management.
  units on a scale | 60 [45 to 70] | 55 [35 to 65] | 60 [40 to 70]
Maintenance (CC SCHFI) [Median (Inter-Quartile Range); unit: units on a scale] — Maintenance is a subscale of the Caregiver Contribution to Self-Care in HF Index (CC SCHFI). The CC-SCHFI is a 22-item scale which measures caregivers' contributions to: HF maintenance, HF management, and HF caregiving self-efficacy (confidence). The maintenance sub-scale ranges from 0-100. Higher scores indicate higher maintenance.
  units on a scale | 86.7 [76.7 to 93.3] | 86.7 [76.7 to 93.3] | 86.7 [76.7 to 93.3]

OUTCOME MEASURES:

1. Primary Outcome: Change in Heart Failure Knowledge
Description: As measured by the Dutch Heart Failure Knowledge Scale, scores range from 0-15; higher scores indicate greater heart failure knowledge.
Time Frame: Baseline (0 days); at follow-up (90 days)
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Enhanced Usual Care | Intervention Arm
Number analyzed (Participants) | 50 | 52
units on a scale | 0.93 [0.05 to 1.81] | 1.88 [1.05 to 2.71]

2. Primary Outcome: Change in Heart Failure Caregiving Self-efficacy
Description: As measured by the Caregiver Contribution to Self-Care in Heart Failure Index, which is a 22-item scale which assesses maintenance, management, and self-efficacy sub-scales separately. Each sub-scale score ranges from 0-100, with greater scores indicating greater contribution to care or self-efficacy.
Time Frame: Baseline (0 days); at follow-up (90 days)
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Enhanced Usual Care | Intervention Arm
Number analyzed (Participants) | 50 | 52
units on a scale | 1.27 [-3.71 to 6.24] | 1.44 [-3.49 to 6.36]

3. Secondary Outcome: Change in Job Satisfaction
Description: As measured by the Work Domain Satisfaction Scale, which is a 5-item scale that measures: 1) job satisfaction among care workers; and 2) examines the associations with work environment factors, work stressors, and health issues. Scores range from 5-20, with higher scores indicating stronger satisfaction.
Time Frame: Baseline (0 days); at follow-up (90 days)
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Enhanced Usual Care | Intervention Arm
Number analyzed (Participants) | 50 | 52
units on a scale | 0.12 [-1.56 to 1.79] | -0.31 [-1.95 to 1.33]

4. Secondary Outcome: Change in Intention to Leave
Description: As measured by the Turnover Intention Scale, which is a 2-item scale that measures workers' intentions of 1) leaving their current job (at their agency) and 2) searching for a new job (in another field) in the next year. ) Responses for both included a 7-point likert scale of: very strongly disagree, strongly disagree, disagree neutral, agree, strongly agree, very strongly agree. Both questions were dichotomized into "agree", "strongly agree", and "very strongly" vs. all other responses.
Time Frame: Baseline (0 days); at follow-up (90 days)
Population: Of the 105 participants that consented to be in the study, 3 participants were lost to follow-up between consents and taking the baseline survey. For non-modeled comparison of count of participants who were thinking of leaving job at 90 days, not all participants responded to the question regarding intentions of 1) leaving their current job and 2) searching for a new job in the baseline survey. Additionally, not all of these participants completed these questions for the 90-day follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care | Intervention Arm
Number analyzed (Participants) | 48 | 50
Participants
  Baseline intention to leave job | 10 | 9
  90 days intention to leave job: number analyzed (Participants) | 36 | 38
  90 days intention to leave job | 6 | 6
  Baseline intention to search for a new job: number analyzed (Participants) | 48 | 49
  Baseline intention to search for a new job | 6 | 5
  90 days intention to search for a new job: number analyzed (Participants) | 35 | 38
  90 days intention to search for a new job | 3 | 3
Statistical Analysis 1: Comparison: Enhanced Usual Care vs Intervention Arm; Outcome measures workers' intentions of leaving their current job. Responses included 7-point likert scale of very strongly disagree-very strongly agree. Dichotomized into "agree", "strongly agree", and "very strongly" vs. other responses. We used logistic mixed regression model to compare outcome between and within study arm. Mixed effects included a variable for time point (baseline/90 days), indicator for study arm, a study arm by time point interaction and subject random intercept; Test type: Equivalence — A p<0.05 considered the threshold for statistical significance; p = 0.974, Regression, Logistic; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.14 to 6.85] — The comparison group is enhanced usual care arm
Statistical Analysis 2: Comparison: Enhanced Usual Care vs Intervention Arm; Outcome measures workers' intentions of searching for a new job. Responses included 7-point likert scale of very strongly disagree-very strongly agree. Dichotomized into "agree", "strongly agree", and "very strongly" vs. other responses. We used logistic mixed regression model to compare outcome between and within study arm. Mixed effects included a variable for time point (baseline/90 days), indicator for study arm, a study arm by time point interaction and subject random intercept; Test type: Equivalence — A p< 0.05 considered the threshold for statistical significance; p = 0.846, Regression, Logistic; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.08 to 7.72] — The comparison group is enhanced usual care arm

5. Other Pre Specified Outcome: Number of Visits to the Emergency Department
Description: All-cause emergency department visits to any emergency department
Time Frame: Baseline (0 days); at follow-up (90 days)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Number of Readmissions to the Hospital
Description: All-cause readmissions to any hospital
Time Frame: Baseline (0 days); at follow-up (90 days)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Preventable 911 Calls
Description: Preventable 911 calls were assessed with 2-close ended questions that we previously used among HHAs: "I have called 911 when that could have been prevented if I had been able to reach my supervisor/the nurse." and "I have called 911 when that could have been prevented if my supervisor and I had been able to reach the client's doctor." Responses for both included a 7-point Likert scale of: very strongly disagree, strongly disagree, disagree neutral, agree, strongly agree, very strongly agree. Both questions dichotomized into "agree", "strongly agree", and "very strongly" vs. all other responses.
Time Frame: Baseline (0 days); at follow-up (90 days)
Population: Of the 105 participants that consented to be in the study, 3 participants were lost to follow-up between consents and taking the baseline survey. For non-modeled comparison of count of participants who were thinking of leaving job at 90 days, not all participants responded to the questions regarding preventable 911 calls in baseline survey. Additionally, not all participants responded to preventable 911 call questions at 90-day follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Usual Care | Intervention Arm
Number analyzed (Participants) | 50 | 52
Participants
  Baseline-preventable 911 call if reached doctor: number analyzed (Participants) | 48 | 51
  Baseline-preventable 911 call if reached doctor | 20 | 26
  90 days-preventable 911 call if reached doctor: number analyzed (Participants) | 37 | 38
  90 days-preventable 911 call if reached doctor | 19 | 13
  Baseline-preventable 911 call if reached nurse/supervisor: number analyzed (Participants) | 49 | 51
  Baseline-preventable 911 call if reached nurse/supervisor | 30 | 28
  90 days-preventable 911 call if reached nurse/supervisor: number analyzed (Participants) | 36 | 38
  90 days-preventable 911 call if reached nurse/supervisor | 18 | 18
Statistical Analysis 1: Comparison: Enhanced Usual Care vs Intervention Arm; Preventable 911 calls if had been able to reach the doctor. Dichotomized into "agree", "strongly agree", and "very strongly" vs. all other responses. We used logistic mixed regression model to compare trajectory of all outcomes between and within study arms. Mixed effects included a fixed effects categorical variable for time point (baseline/90days), and indicator for study arm (enhanced usual care/intervention), a study arm by time point interaction and subject specific random intercept; Test type: Equivalence — A p<0.05 was considered the threshold for statistical significance; p = 0.043, Regression, Logistic; Odds Ratio (OR) = 0.18, 95% CI 2-sided [0.03 to 0.94] — The comparison group is enhanced usual care arm
Statistical Analysis 2: Comparison: Enhanced Usual Care vs Intervention Arm; Preventable 911 calls if had been able to reach the nurse/supervisor. Dichotomized into "agree", "strongly agree", and "very strongly" vs. other responses. We used logistic mixed regression model to compare trajectory of all outcomes between and within study arms. Mixed effects included a fixed effects categorical variable for time point (baseline/90days), and indicator for study arm (enhanced usual care/intervention), a study arm by time point interaction and subject specific random intercept; Test type: Equivalence — A p<0.05 considered the threshold for statistical significance; p = 0.99, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.22 to 4.58]

ADVERSE EVENTS:
Time Frame: 90 days from baseline survey
Description: Of the 105 participants that consented to be in the study, 3 participants were lost to follow-up between consents and taking the baseline survey.
Arm/Group | Enhanced Usual Care | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/52
Other Adverse Events (participants affected / at risk) | 0/50 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT04239911/Prot_SAP_ICF_001.pdf